CLINICAL TRIAL: NCT02443454
Title: Short and Long-term Results of Arterial Stiffness and Central Aortic Pressure After Kidney Transplantation
Acronym: PWV/CP/KTx
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Łukasz Czyżewski, Łukasz Czyżewski, Medical University of Warsaw
Other Study IDs: PWV/CP/KTx/2015/05
Record Dates: First submitted 2015-05-10; First posted 2015-05-13 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Arterial Calcification; Aortic Stiffness; High Blood Pressure (& [Essential Hypertension])
MeSH Terms: conditions — Hypertension; Essential Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients after kidney transplantation: Short and Long-term results containing first 10 years after KTx.
  Interventions: Device: Device: Complior Analyse System; Device: Tanita BC 418- Bioelectrical impedance analysis
- Healthy subjects: Medical staff: medical doctors, nurses
  Interventions: Device: Device: Complior Analyse System

INTERVENTIONS:
Device: Device: Complior Analyse System — Monitoring of Arterial Stiffness and Central Aortic Pressure
Device: Tanita BC 418- Bioelectrical impedance analysis — The device measured the size of total body water (TBW), fat mass (FM%), visceral fat%, fat free mass (FFM), and basal metabolic rate (BMR) (kcal).
  Groups: Patients after kidney transplantation

SUMMARY:
Central blood pressure and pulse wave velocity were measured using a Complior Analyse device in Short and Long-term after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* functioning graft longer than 3 months to 10 years
* no clinical cardiovascular disease during the 6 months preceding entry
* stable graft function- glomerular filtration rate > 30 ml/min/1.73 m2, creatinine concentration <2.5 mg/dl
* medical staff (medical doctors, nurses)

Exclusion Criteria:

* not meet the above criteria
* episode of illness (for example: infection)
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 100 consecutive patients admitted to routine visin in Transplant Centre and 30 healthy subjects were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Differences in carotid-femoral pulse wave velocity [m/s] in short and long-term postoperative period. | 1 day
  Measurements will be performed in routine visits in Transplant Centre.

SECONDARY OUTCOMES:
Differences in central aortic pressure [mmHg] in short and long-term postoperative period. | 1 day
  Measurements will be performed in routine visits in Transplant Centre.
Differences in central aortic pressure [mmHg] and cuff blood pressure [mmHg] in short and long-term postoperative period. | 1 day
  Measurements will be performed in routine visits in Transplant Centre.

CONTACTS AND LOCATIONS:
Overall Officials: Łukasz Czyżewski, PhD, Study Chair — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Warsaw, Mazovian, Poland

REFERENCES:
- [Background] Czyzewski L, Sanko-Resmer J, Wyzgal J, Kurowski A. Comparative analysis of hypertension and its causes among renal replacement therapy patients. Ann Transplant. 2014 Nov 3;19:556-68. doi: 10.12659/AOT.891248. PMID 25365639
- [Background] Czyzewski L, Wyzgal J, Kolek A. Evaluation of selected risk factors of cardiovascular diseases among patients after kidney transplantation, with particular focus on the role of 24-hour automatic blood pressure measurement in the diagnosis of hypertension: an introductory report. Ann Transplant. 2014 Apr 28;19:188-98. doi: 10.12659/AOT.890189. PMID 24770703
- [Background] Czyzewski L, Sanko-Resmer J, Wyzgal J, Kurowski A. Assessment of health-related quality of life of patients after kidney transplantation in comparison with hemodialysis and peritoneal dialysis. Ann Transplant. 2014 Nov 9;19:576-85. doi: 10.12659/AOT.891265. PMID 25382249